CLINICAL TRIAL: NCT07374588
Title: The Effect of Medication Education on Treatment Adherence and Side Effects in Psychiatric Inpatients: An Intervention Study
Brief Title: Impact of Medication Education on Adherence and Side Effects
Acronym: MED-ADHERE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, özge kısaoğlu, Associate Professor of Psychiatric Nursing, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-07/33
Record Dates: First submitted 2026-01-10; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder With Psychotic Features; Major Depressive Disorder With Psychotic Features
Keywords: Medication Education; Psychiatric Inpatients; Psychoeducation; Treatment Adherence; Medication Side Effects
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Treatment Adherence and Compliance; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either an intervention group receiving structured medication education in addition to routine care or a control group receiving routine psychiatric inpatient care alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medication Education + Routine Care (Experimental): Participants in this arm will receive routine psychiatric inpatient care in addition to a structured medication education program. The medication education aims to improve medication adherence and enhance coping with medication-related side effects. The education will be delivered by the researchers in two sessions, each lasting 45 minutes, using teaching, discussion, and role-playing methods.
  Interventions: Behavioral: Medication Education Program
- Routine Care (Active Comparator): Participants in this arm will receive routine psychiatric inpatient care only, including standard pharmacological treatment and nursing care provided according to hospital protocols. No additional medication education will be provided.
  Interventions: Behavioral: Routine Psychiatric Inpatient Care

INTERVENTIONS:
Behavioral: Medication Education Program — Structured medication education provided in addition to routine psychiatric inpatient care.
  Arms: Medication Education + Routine Care
Behavioral: Routine Psychiatric Inpatient Care — Standard psychiatric inpatient care including pharmacological treatment and routine nursing care provided according to hospital protocols. No additional medication education is provided.
  Arms: Routine Care

SUMMARY:
Severe mental disorders such as schizophrenia, bipolar disorder, and psychotic depression often require long-term or lifelong medication treatment. However, many psychiatric patients have difficulty adhering to their prescribed medication regimens due to factors such as lack of information, fear of side effects, and negative experiences with psychotropic medications. Poor treatment adherence is associated with symptom relapse, prolonged hospitalization, increased rehospitalization rates, reduced quality of life, and higher health care costs.

Medication education is a key psychosocial intervention aimed at improving patients' understanding of their illness, treatment process, and potential medication side effects. Providing structured medication education may enhance treatment adherence and help patients recognize and manage side effects more effectively.

This intervention study aims to evaluate the effect of a structured medication education program on treatment adherence and medication-related side effects among psychotic inpatients hospitalized in a psychiatric clinic, including patients diagnosed with schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar disorder with psychotic features, and major depressive disorder with psychotic features. The findings of this study are expected to contribute to the development of effective psychosocial interventions to improve medication adherence and treatment outcomes in psychiatric inpatient settings.

DETAILED DESCRIPTION:
Mental disorders with psychotic features, such as schizophrenia, schizoaffective disorder, bipolar disorder with psychotic features, and psychotic depression, are chronic conditions that often require long-term or lifelong pharmacological treatment. Despite the effectiveness of psychotropic medications in symptom control and relapse prevention, treatment non-adherence remains a major challenge in psychiatric care. Medication non-adherence in psychiatric patients is associated with increased relapse rates, prolonged hospitalization, involuntary admissions, poorer prognosis, increased suicide risk, and higher health care costs. One of the most frequently reported reasons for non-adherence is the experience of, or fear of experiencing, medication-related side effects.

Medication education is a structured psychosocial intervention designed to improve patients' knowledge about their illness, prescribed medications, expected benefits, possible side effects, and strategies for managing adverse effects. Increasing patients' understanding of their treatment may enhance insight, reduce anxiety related to medication use, and improve treatment adherence.

This intervention study aims to evaluate the effect of a structured medication education program on treatment adherence and medication-related side effects among psychotic inpatients hospitalized in a psychiatric clinic. The study population consists of patients diagnosed with schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar disorder with psychotic features, and major depressive disorder with psychotic features.

Participants will receive routine psychiatric inpatient care. In addition, the intervention group will receive a structured medication education program delivered by trained mental health professionals. The medication education program includes information about the nature of the psychiatric illness, the purpose and benefits of prescribed medications, correct medication use, potential side effects, and strategies for recognizing and managing common adverse effects. Educational sessions are designed to be interactive and tailored to patients' cognitive and clinical status.

Treatment adherence and medication-related side effects will be assessed using validated measurement tools at predefined time points. The outcomes of the intervention group will be compared with those of the control group receiving standard care alone.

The results of this study are expected to provide evidence on the effectiveness of medication education as a psychosocial intervention for improving treatment adherence and reducing the negative impact of medication side effects in psychiatric inpatient settings. The findings may contribute to the development of standardized educational interventions aimed at improving long-term treatment outcomes and quality of life in patients with severe mental disorders.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Hospitalized in a psychiatric inpatient clinic
* Diagnosed with schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar disorder with psychotic features, or major depressive disorder with psychotic features
* Receiving psychotropic medication treatment
* Clinically stable and able to participate in educational sessions
* Able to communicate verbally and understand the content of the education
* Provided written informed consent

Exclusion Criteria:

* Presence of severe cognitive impairment or intellectual disability
* Acute medical or neurological conditions that may interfere with participation
* Severe agitation or acute psychotic symptoms preventing participation
* Hearing or communication impairments that limit participation in educational sessions
* Participation in another psychosocial intervention study during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Treatment Adherence | Baseline and at the end of the intervention period during hospitalization (up to 5 days)
  Treatment adherence will be assessed by evaluating patients' adherence to prescribed psychotropic medications, including regular medication use and compliance with the treatment regimen, using a validated medication adherence assessment tool.

SECONDARY OUTCOMES:
Medication-Related Side Effects | Baseline and at the end of the intervention period during hospitalization (up to 5 days)
  Medication-related side effects will be assessed by evaluating the presence, frequency, and severity of psychotropic medication side effects using a validated side effect assessment scale.

IPD SHARING:
Plan to Share IPD: No